CLINICAL TRIAL: NCT00770354
Title: A Phase II, Randomised, Open-Label, Multicentre Study of AS1402 in Combination With Letrozole as First Line Treatment in Postmenopausal Women With Locally Advanced or Metastatic Breast Cancer
Brief Title: Phase II Study of AS1402 Combined With Letrozole to Treat Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Antisoma Research (Industry)
Responsible Party: Gary Acton, Antisoma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1402-C-201
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Breast Carcinoma
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — epitumomab; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): AS1402 plus letrozole
  Interventions: Drug: AS1402
- 2 (Active Comparator): Letrozole
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: AS1402 — A complete treatment cycle spans 28 days. Patients randomised to AS1402 will receive a 1-hour infusion of 9 mg/kg on day 1, 8, 15 and 22 of each cycle. Patients will receive letrozole (2.5 mg daily tablet).
  Other Names: huHMFG1
  Arms: 1
Drug: Letrozole — Daily 2.5 mg oral letrozole tablet
  Other Names: Femara
  Arms: 2

SUMMARY:
The aim of this study is to compare the overall tumour response rate per RECIST in postmenopausal women with metastatic or locally advanced breast cancer receiving AS1402 in combination with letrozole compared to letrozole alone

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic breast cancer not amenable to curative therapy
* Measurable disease according to the RECIST criteria
* Documented estrogen receptor-positive and/or progesterone receptor-positive tumour
* Postmenopausal women

Exclusion Criteria:

* Prior chemotherapy and/or endocrine therapy for advanced breast disease
* Relapse within 12 months after treatment discontinuation of an aromatase inhibitor in the adjuvant setting
* Unknown hormonal receptor status
* Known HER2/neu-positivity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is overall response rate (ORR) | Radiological evaluations are performed every 12 weeks up to progression

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Radiological evaluations are performed every 12 weeks up to progression
Time to progression (TTP) | Radiological evaluations are performed every 12 weeks up to progression
Duration of overall response and duration of stable disease | Radiological evaluations are performed every 12 weeks up to progression
Clinical benefit rate (CBR) | Radiological evaluations are performed every 12 weeks up to progression
Safety and tolerability of AS1402 when combined with letrozole | Radiological evaluations are performed every 12 weeks up to progression

CONTACTS AND LOCATIONS:
Overall Officials: Gary Acton, MA MBBS MRCP, Study Director — Antisoma Research; Nuhad K Ibrahim, MD FACP, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- Russia (2):
  - State Medical Institution, Pyatigorsk, Stavropol Kray
  - State Therapeutical and Prophylactic Institution: Chelyabinsk Regional Oncological Center, Chelyabinsk

REFERENCES:
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562
- [Derived] Ibrahim NK, Yariz KO, Bondarenko I, Manikhas A, Semiglazov V, Alyasova A, Komisarenko V, Shparyk Y, Murray JL, Jones D, Senderovich S, Chau A, Erlandsson F, Acton G, Pegram M. Randomized phase II trial of letrozole plus anti-MUC1 antibody AS1402 in hormone receptor-positive locally advanced or metastatic breast cancer. Clin Cancer Res. 2011 Nov 1;17(21):6822-30. doi: 10.1158/1078-0432.CCR-11-1151. Epub 2011 Aug 30. PMID 21878535